CLINICAL TRIAL: NCT02225171
Title: Physicians' Experiences With and Attitudes Toward Non-Medical Sex Selection Through Preimplantation Genetic Diagnosis
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914166; 14-HG-N166
Record Dates: First submitted 2014-08-23; First posted 2014-08-26 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Genetics; Attitudes
Keywords: Assisted Reproductive Technology; Behavior; Health Care Provider; Ethical Concerns; Decision Making; Natural History
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians: 15 physicians each will be interviewed from the specialties of reproductive endocrinology and obstetrics/gynecology.

SUMMARY:
Preimplantation genetic diagnosis (PGD) is an assisted reproductive technology (ART) by which embryos, created through in vitro fertilization (IVF), can be screened for genetic conditions or traits before they are implanted into a woman s uterus. Within the past few years, a controversial non-medical use of PGD has gained recognition as having possible significant ethical implications. Non-medical sex selection (NMSS) describes the use of PGD technology to choose the sex of a child for social, as opposed to medical, reasons. In the US and a select few other countries, it is legal to use NMSS for family balancing, or the intentional selection of an underrepresented sex to balance a family where the majority of the children are of one sex. Proponents of family balancing believe that NMSS is an expression of reproductive autonomy and is ethically acceptable on those grounds. Opponents are more likely to cite beneficence (toward the existing children and the potential future child) and justice (resource allocation and access, for example) as the basis for concerns around NMSS and family balancing specifically. In the US and other countries, healthcare providers (HCPs) are often the gatekeepers to this technology. There is little research exploring the experiences of HCPs with PGD and NMSS. The Moral Experience framework (Hunt and Carnevale, 2011) is useful for understanding the potential concerns of HCPs as well as their feelings and behaviors evoked by lived and hypothetical experiences around NMSS. Also of interest is how HCPs feel that decisions about NMSS are made and their preferences as to how they should be made. Finally, there is concern that NMSS may be the first in a line of non-medical uses for PGD and that a slippery slope toward what some describe as designer babies will follow. We are interested in eliciting the traits that HCPs believe are hypothetically appropriate or inappropriate for PGD and how they make the distinction. Interviews with HCPs (OBGYNs and reproductive endocrinologists) on these topics will be transcribed and subjected to thematic analysis in order to identify common themes. An understanding of the experiences and attitudes of this stakeholder population can help clarify current issues at individual, societal, and global levels and future directions for research and policy....

DETAILED DESCRIPTION:
Preimplantation genetic diagnosis (PGD) is an assisted reproductive technology (ART) by which embryos, created through in vitro fertilization (IVF), can be screened for genetic conditions or traits before they are implanted into a woman s uterus. Within the past few years, a controversial non-medical use of PGD has gained recognition as having possible significant ethical implications. Non-medical sex selection (NMSS) describes the use of PGD technology to choose the sex of a child for social, as opposed to medical, reasons. In the US and a select few other countries, it is legal to use NMSS for family balancing, or the intentional selection of an underrepresented sex to balance a family where the majority of the children are of one sex. Proponents of family balancing believe that NMSS is an expression of reproductive autonomy and is ethically acceptable on those grounds. Opponents are more likely to cite beneficence (toward the existing children and the potential future child) and justice (resource allocation and access, for example) as the basis for concerns around NMSS and family balancing specifically. In the US and other countries, healthcare providers (HCPs) are often the gatekeepers to this technology. There is little research exploring the experiences of HCPs with PGD and NMSS. The Moral Experience framework (Hunt and Carnevale, 2011) is useful for understanding the potential concerns of HCPs as well as their feelings and behaviors evoked by lived and hypothetical experiences around NMSS. Also of interest is how HCPs feel that decisions about NMSS are made and their preferences as to how they should be made. Finally, there is concern that NMSS may be the first in a line of non-medical uses for PGD and that a slippery slope toward what some describe as designer babies will follow. We are interested in eliciting the traits that HCPs believe are hypothetically appropriate or inappropriate for PGD and how they make the distinction. Interviews with HCPs (OBGYNs and reproductive endocrinologists) on these topics will be transcribed and subjected to thematic analysis in order to identify common themes. An understanding of the experiences and attitudes of this stakeholder population can help clarify current issues at individual, societal, and global levels and future directions for research and policy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must:

* speak English
* be at least 18 years of age
* currently be practicing in a clinical setting in the US
* have familiarity with PGD i.e. have discussed PGD with a patient or colleague in any context

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 physicians each will be interviewed from the specialties of reproductive endocrinology and obstetrics/gynecology.@@@
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2014-08-23 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Experiences | Enrollment
  This study seeks to describe the experiences of healthcare providers around pre- implantation genetic diagnosis (PGD) for non-medical sex selection (NMSS), with a particular focus on potential ethical concerns, their role in the decision-making process, and their views on future appropriate and inappropriate non-medical uses of PGD.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erby, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States